CLINICAL TRIAL: NCT06857851
Title: Optimizing Deep Brain Stimulation to Improve Visuomotor Function in Parkinson's Disease
Acronym: DBS strabismus
Status: Not yet recruiting | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: C5298-R; I01RX005298-01A1 (NIH)
Record Dates: First submitted 2025-02-19; First posted 2025-03-04 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Deep brain stimulation; subthalamic nucleus
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Parkinson's disease with DBS: This is the only group. The patients in this group will have bilateral subthalamic region deep brain stimulator. They will be recruited after they are therapeutically optimized on stimulation as well as medical therapy.

SUMMARY:
Inability to align and refocus the eyes on the objects at different depths, i.e., vergence impairment and strabismus, frequently affects the quality of life in patients with Parkinson's disease. The investigators study aims to understand the location-specific effects of subthalamic region deep brain stimulation on vergence and strabismus by integrating the patient-specific deep brain stimulation models and high-resolution eye-tracking measures. The knowledge gained will allow the investigators to find the most beneficial stimulation location and parameters for improving binocular coordination, strabismus, and vergence while preserving the ability to treat motor symptoms in Parkinson's disease.

DETAILED DESCRIPTION:
The victims of very common condition Parkinson's disease (PD) are known to have tremor, rigidity, and slow movements. PD, in addition to its effects on human movements, also affects many other aspect of the brain's function. Impairment of vision is frequently seen in PD. These patients have difficulties with holding their eyes steady at a given point, seamlessly look around and read, and refocus their eyes from one image to the other while looking at objects that are at different depths. About third of the PD patients have problems coordinating the movement of two eyes together, i.e., abnormal vergence and strabismus. Latter results in disabling double vision and abnormal depth perception. Most treatment options available to PD patients are limited to their effects on tremor, stiffness, and slowness - their effects on visual function is very limited. Eye surgeries are not ideal treatment strategies for these conditions given constantly changing state of the PD brain due to its degenerative nature. Cutting edge deep brain stimulation (DBS) surgery has variable effects on the eye movements and vergence function and strabismus in PD. The goal of the investigators research program is to identify the best possible therapeutic strategy using DBS to improve vergence eye movements and strabismus in PD while continuing to offer its other benefits. The investigators multidisciplinary program has two aspects. One part of the study will examine the effects of DBS on vergence abnormalities and strabismus affecting their ability to focus at various depths. Using state of art, high-resolution, research grade ophthalmic equipment the investigators will examine fine details of how DBS alters the patients' ability to refocus and how it changes the alignment between the two eyes that can cause double vision and abnormal depth perception. Once the investigators identify these characteristic changes, the investigators will correlate them with the stimulated anatomical location within the same patient's brain determined using combination of novel computer simulations of DBS and the patient's own MRI. The knowledge gained will allow the investigators to find the ideal stimulation locations that is most beneficial to the patient for improvement in vision while continuing to offer benefits for tremor, rigidity, and slow movements.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson's disease with bilateral STN DBS
* Availability of pre-operative MR images (with a T1-weighted, gradient-echo sequence) and ability to get post-operative MRI or CT scans
* Hoehn and Yahr stage 2-4 when off medication, and a stable antiparkinsonian medication regimen and DBS parameter settings

Exclusion Criteria:

* Previous surgical therapy for Parkinson's disease (other than DBS)
* Dementia
* Clinically significant untreated depression or anxiety
* Clinical features suggestive of atypical parkinsonism

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: United States Military Veterans
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Eye alignment - vergence gain | One month
  The investigators will measure vergence gain as one outcome measure. This measure will be calculated by measuring ratio of observed versus expected difference between the horizontal angular positions of the right and left eye as participants move gaze from far to near or vice versa.
Strabismus | One month
  The investigators will measure difference in position of right versus left eye as participants hold gaze on object of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Aasef G. Shaikh, MD PhD, Principal Investigator — Louis Stokes VA Medical Center, Cleveland, OH
Locations (1):
- Louis Stokes VA Medical Center, Cleveland, OH, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No